CLINICAL TRIAL: NCT04745325
Title: Assessing the Effectiveness and Mechanisms of Action of a Smartphone App Designed to Reduce Unhealthy Alcohol Consumption: Randomized Controlled Trial
Brief Title: Randomized Trial of a Smartphone App Designed to Reduce Unhealthy Alcohol Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 052/2020
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone app - full access (Experimental): A smartphone app containing 5 modules: 1) personalized feedback on alcohol use (containing normative feedback by age and sex for those located in the Canada), 2) self-monitoring and goal setting tool, 3) tool to choose a designated driver, 4) blood alcohol content (BAC) calculator, and 5) educational information on alcohol use and its consequences (i.e. "fact sheets").
  Interventions: Behavioral: SMAART Canada smartphone app
- Smartphone App - education only (Active Comparator): A version of the Smartphone app containing only the module with the educational information on alcohol use and its consequences (i.e. "fact sheets").
  Interventions: Behavioral: SMAART Canada smartphone app

INTERVENTIONS:
Behavioral: SMAART Canada smartphone app — a smartphone app designed to promote reductions in alcohol consumption among people who drink in a hazardous fashion

SUMMARY:
Smartphone apps targeting alcohol consumption are increasingly employed as a means to help people reduce their alcohol consumption. Recognizing this potential, there has been an explosion of app development for unhealthy alcohol use, as well as other health-related behaviours. This study will recruit people who consume alcohol in an unhealthy manner. Participants will be assigned by chance to one of two groups and will be contacted 6 months after consenting to the study to assess changes in their drinking. In addition, this study will help us understand which components of the smartphone app are important to use in order to promote reductions in alcohol consumption. An app with proven efficacy, made widely available and free-of-charge to Canadians, will provide a much needed option to help those in need to reduce their alcohol use.

DETAILED DESCRIPTION:
Unhealthy alcohol use is common and causes tremendous harm. Most people with unhealthy alcohol use will never seek formal alcohol treatment. As an alternative, smartphone apps have been developed as one means to provide help to people concerned about their alcohol use. While such apps are widely available, the large majority have little or no evidence base, and research has indicated that some may actually do more harm than good. An app with proven efficacy at reducing alcohol consumption is needed in order to capitalize on this opportunity to motivate the large number of people seeking assistance using this promising technology.

This study will recruit people who consume alcohol in an unhealthy manner. Participants will be assigned by chance to one of two groups to either receive access to: 1) the full app; or 2) a copy of the app where only the educational content is provided (as opposed to the full intervention content of the app). Participants will be contacted 6 months after consenting to the study to assess changes in their drinking. We predict that the full app will lead to larger reductions in drinking and a more sustained impact than the educational content only app. In addition, this study will help us understand which components of the smartphone app are important to use in order to promote reductions in alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* score of 8 or more on the Alcohol Use Disorders Identification Test
* currently us a smartphone running iOS or Android

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Total number of drinks consumed in a typical week | 6-months follow-up
  self-reported change

SECONDARY OUTCOMES:
Frequency of heavy drinking days | 6-months follow-up
  self-reported change
Number of consequences associated with drinking | 6-months follow-up
  self-reported change

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Canada

REFERENCES:
- [Derived] Cunningham JA, Godinho A, Schell C, Studer J, Wardell JD, Garnett C, Bertholet N. Randomized controlled trial of a smartphone app designed to reduce unhealthy alcohol consumption. Internet Interv. 2024 May 17;36:100747. doi: 10.1016/j.invent.2024.100747. eCollection 2024 Jun. PMID 38812955